CLINICAL TRIAL: NCT00002093
Title: A Randomized Phase III Clinical Trial of Daunoxome Versus Combination Chemotherapy With Adriamycin/Bleomycin/Vincristine (ABV) in the Treatment of HIV-Associated Kaposi's Sarcoma.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nexstar Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 121A; 103-09
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-03

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Vincristine; Sarcoma, Kaposi; Liposomes; Doxorubicin; Acquired Immunodeficiency Syndrome; Bleomycin; Daunorubicin; Drug Carriers
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Daunorubicin; Bleomycin; Vincristine; Doxorubicin

INTERVENTIONS:
Drug: Daunorubicin (liposomal)
Drug: Bleomycin sulfate
Drug: Vincristine sulfate
Drug: Doxorubicin hydrochloride

SUMMARY:
To compare the toxicity profiles (severity and time to onset from initiation of therapy) between daunorubicin (liposomal) and combination chemotherapy with doxorubicin/bleomycin/vincristine (ABV), with both regimens administered in combination with antiretroviral therapy. To compare the duration of responses, response rates, and times to response.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* Advanced Kaposi's sarcoma.

Prior Medication:

Allowed:

* Prior intralesional vinblastine.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Acute intercurrent infection other than genital herpes.
* Uncompensated cardiovascular, hepatic, renal, or pulmonary disease unrelated to Kaposi's sarcoma.
* Symptomatic peripheral neuropathy.
* Any condition that compromises ability to give informed consent or complete the study.

Concurrent Medication:

Excluded:

* Concurrent ganciclovir.

Patients with the following prior conditions are excluded:

* Symptomatic AIDS-defining opportunistic infection within 2 weeks of entry.
* History of malignancy other than Kaposi's sarcoma, basal cell carcinoma, or carcinoma in situ of the cervix.

Prior Medication:

Excluded:

* Prior systemic chemotherapy.
* Intralesional therapies within 7 days prior to study entry.
* Growth factors (G-CSF or GM-CSF), immune modifiers, or investigational agents within 14 days prior to study entry.
* Interferon preparations (alpha or beta) within 28 days prior to study entry.

Prior Treatment:

Excluded within 7 days prior to study entry:

* Radiation.
* Local therapies (e.g., cryotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Univ of Arizona / Arizona Cancer Ctr, Tucson, Arizona
  - Kenneth Norris Jr Cancer Hosp, Los Angeles, California
  - Desert Hosp Comprehensive Cancer Ctr, Palm Springs, California
  - Saint Francis Mem Hosp, San Francisco, California
  - Davies Med Ctr, San Francisco, California
  - Denver Gen Hosp, Denver, Colorado
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Miami Dept of Medicine, Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - New England Deaconess Hosp, Boston, Massachusetts
  - New York Univ Med Ctr, New York, New York
  - Kaiser Permanente Med Ctr, Portland, Oregon
  - Dr Edward Stool, Houston, Texas

REFERENCES:
- [Background] Gill PS, Wernz J, Scadden DT, Cohen P, Mukwaya GM, von Roenn JH, Jacobs M, Kempin S, Silverberg I, Gonzales G, Rarick MU, Myers AM, Shepherd F, Sawka C, Pike MC, Ross ME. Randomized phase III trial of liposomal daunorubicin versus doxorubicin, bleomycin, and vincristine in AIDS-related Kaposi's sarcoma. J Clin Oncol. 1996 Aug;14(8):2353-64. doi: 10.1200/JCO.1996.14.8.2353. PMID 8708728
- [Background] Savage GE, Gable C, Motte K, Dixon C, Becker R. A pharmacoeconomic analysis of Kaposi's sarcoma patients based on a clinical trial of ABV vs. DaunoXome. Int Conf AIDS. 1996 Jul 7-12;11(Program Supplement):32 (abstract no LBB6048)